CLINICAL TRIAL: NCT04406610
Title: Chimeric Antigen Receptor-Modified T Cells for GD2 Positive Recurrent and Metastatic Glioma
Brief Title: CAR-T Cell Immunotherapy for GD2 Positive Glioma Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Project terminated due to revision of local regulations
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAR-T
Record Dates: First submitted 2019-09-10; First posted 2020-05-28 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Glioma of Brain; CAR-T Cell Immunotherapy
Keywords: CAR-T cell immunotherapy; GD2; glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GD2 CAR-T (Experimental): Treated by GD2 CAR-T therapy intravenously
  Interventions: Biological: GD2 CAR-T immunotherapy
- Control (No Intervention): With no medical intervention

INTERVENTIONS:
Biological: GD2 CAR-T immunotherapy — Antigen-specific T cell therapy
  Other Names: CAR-T for glioma
  Arms: GD2 CAR-T

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CAR-T cell immunotherapy in treating with GD2 positive glioma patients.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) is a recombinant receptor with both antigen-binding and T cell activating functions. Chimeric antigen receptor T cell Immunotherapy has more advantages compared with conventional immunotherapy, especially in dealing with patients of hematologic malignancies and solid malignant tumors.This study design a novel specific Chimeric antigen receptor aiming at GD2 antigen.After CAR-T cell infusion,At periodic intervals, the investigators will evaluate clinical symptoms Improved conditions of this disease.Through this study,the investigators will evaluate the safty and effectiveness of CAR-T cell immunotherapy in treating with GD2 positive glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 2 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
Classification of adverse reactions | 3 months
  To observe the common 1-4 levels of side effects

SECONDARY OUTCOMES:
Progression free survival （PFS）of patients | 1 year
  PFS was defined as the interval between treatment initiation and local relapse, distant metastasis, or death, whichever occurred first.